CLINICAL TRIAL: NCT03507803
Title: Effects of Gait Biofeedback and Impairment-based Rehabilitation in Individuals With Chronic Ankle Instability
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Virginia (Other)
Responsible Party: Principal Investigator, Jay Hertel, PhD, ATC, Principal Investigator, University of Virginia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 20446
Record Dates: First submitted 2018-02-15; First posted 2018-04-25 (Actual); Last update posted 2018-05-16 (Actual); Status verified 2018-05

CONDITIONS: Ankle Sprains; Ankle Injuries
Keywords: Gait training; Walking
MeSH Terms: conditions — Ankle Injuries

STUDY DESIGN:
Intervention Model Description: Participants will be randomized at the baseline visit to either the intervention or control group. The intervention group will receive gait biofeedback. Participants will remain within their designated allocation for the entire study.
Who Masked: Care Provider
Masking Description: Clinician involved in rehabilitation will not know if participant has been enrolled in the gait biofeedback arm or the control (no biofeedback) arm.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Gait Biofeedback (Experimental): This group will receive audiovisual feedback about the position of their foot during walking. Feedback will be provided over 8 total sessions.
  Interventions: Other: Gait Biofeedback
- Control (No Intervention): This arm will not receive any audiovisual feedback about the position of their foot during walking.

INTERVENTIONS:
Other: Gait Biofeedback — Feedback will appear on screen in front of participants during walking. If their foot is too inverted (determined by researcher) the object on the screen will turn red and an audio tone will be heard. If the participant corrects the foot position, the object will turn green and the audio tone will not be heard.
  Arms: Gait Biofeedback

SUMMARY:
Individuals with chronic ankle instability (CAI) have demonstrated altered gait patterns. Gait training may be necessary to address these alterations as protocols focusing solely on strength or balance have not been shown to impact walking gait. Biofeedback about the foot position during walking may help improve gait biomechanics. The purpose is to determine whether a 4-week rehabilitation program that includes biofeedback has beneficial effects on self-reported function and ankle gait kinematics compared to rehabilitation alone in people with CAI. The design is a single-blinded randomized controlled trial. Participants will complete baseline self-reported function questionnaires and walking gait trials and then be randomized to complete 4- weeks of supervised rehabilitation with or without audiovisual biofeedback. Follow up emails will ask for participant information about ankle health and to complete questionnaires about their ankle for 6 months and 12 months after completing rehabilitation.

DETAILED DESCRIPTION:
This study will require 10 visits for all participants. Both groups will participate in baseline and follow-up gait assessments involving walking on a treadmill at 1.34 m/s. Follow-up visits will be conducted within 72 hours of the participant's final rehabilitation session. Using a rigid cluster marker setup, reflective markers will be placed on the upper back, sacrum, and bilaterally on the thigh, shank, rearfoot, and forefoot. A 5-minute familiarization period will be completed to ensure participants are comfortable and walking as normally as possible. Following the familiarization period, 1-minute of continuous gait data will be collected. The data collected during baseline and follow-up gait assessments will be used to analyze the primary and secondary outcome measures for kinematics. Participants will also complete the patient reported outcomes (FAAM ADL & Sport Subscale) at the baseline and follow-up visits.

Impairment-based Rehabilitation:

Four weeks of supervised rehabilitation (8 sessions) will be provided to both groups. This rehabilitation paradigm has been previously reported by Donovan and Hertel. Impairment-based rehabilitation involves identifying and treating deficits in 4 broad domains including range of motion (ROM), strength, balance, and functional exercises by using an "asses, treat, re-assess" approach. Previously reported intervention methods will be used in this study. The clinician administering the rehabilitation will be blinded to the subjects' intervention group status.

Intervention:

Gait training using visual feedback for frontal plane ankle position at initial contact (IC) will be projected onto a screen in front of the treadmill.

Gait Training Protocol:

The goal of this protocol is to improve the position of the ankle at IC using visual feedback gait training over the course of 4 weeks. The intervention group will participate in 2 sessions of gait training per week for 4 weeks using intermittent feedback described by Noehren et al. The Motion Monitor is a software system uses body movements to provide visual feedback to the participant by using information from retroreflective markers on the body that are captured by the cameras. The software will use the position of the rearfoot marker cluster in relation to the shank marker cluster to determine the rearfoot inversion angle at IC and provide visual biofeedback information for the next step. Visual feedback in the shape of a line will be displayed as an image projected onto a screen in front of the treadmill representing frontal plane inversion angle. The line will adjust (similar to a teeter-totter) according to the position of the foot and will change color accordingly. When the ankle position is too inverted, the line will turn red and an audio tone will be heard by the participant. When the ankle position is in a good position, the line will turn green and the tone will not be heard.

ELIGIBILITY:
Inclusion Criteria:

* >1 Ankle Sprain (>12 months prior)
* Physically active (>1.5 hr/week)
* > 10 on Identification of Functional Ankle Instability (IdFAI)
* < 90 Foot and Ankle Ability Measure (FAAM) Activities of Daily Living (ADL)
* < 85 FAAM Sport

Exclusion Criteria:

* Hx of LE fracture
* Hx of LE surgery
* Hx of ankle sprain within last 6 weeks
* Participating in physical therapy for ankle
* Multiple Sclerosis
* Marfan's Syndrome
* Lumbosacral Radiculopathy
* Ehlers-Danlos Syndrome
* Diabetes Mellitus
* Pregnant (self-reported)
* Unable to provide informed consent

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2018-02-15 (Actual); Primary Completion 2019-03 (Estimated); Study Completion 2020-03 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline Ankle Frontal Plane Angle During Gait | Baseline, 4 weeks
  Ankle frontal plane angle will be assessed throughout the gait cycle using ensemble curves analysis.

SECONDARY OUTCOMES:
Change from Baseline Ankle Sagittal Plane Angle During Gait | Baseline, 4 weeks
  Ankle sagittal plane angle will be assessed throughout the gait cycle using ensemble curves analysis.
Change from Baseline Ankle Transverse Plane Angle During Gait | Baseline, 4 weeks
  Ankle transverse plane angle will be assessed throughout the gait cycle using ensemble curves analysis.
Change from Baseline Hip Frontal Plane Angle During Gait | Baseline, 4 weeks
  Hip frontal plane angle will be assessed throughout the gait cycle using ensemble curves analysis.
Change from Baseline Hip Sagittal Plane Angle During Gait | Baseline, 4 weeks
  Hip sagittal plane angle will be assessed throughout the gait cycle using ensemble curves analysis.
Change from Baseline Hip Transverse Plane Angle During Gait | Baseline, 4 weeks
  Hip transverse plane angle will be assessed throughout the gait cycle using ensemble curves analysis.
Change from Baseline Knee Frontal Plane Angle During Gait | Baseline, 4 weeks
  Knee frontal plane angle will be assessed throughout the gait cycle using ensemble curves analysis.
Change from Baseline Knee Sagittal Plane Angle During Gait | Baseline, 4 weeks
  Knee sagittal plane angle will be assessed throughout the gait cycle using ensemble curves analysis.
Change from Baseline Knee Transverse Plane Angle During Gait | Baseline, 4 weeks
  Knee transverse plane angle will be assessed throughout the gait cycle using ensemble curves analysis.
Change from Baseline Range of motion | Baseline, 4 weeks
  Ankle range of motion will be assessed using a plastic goniometer
Change from Baseline Balance | Baseline, 4 weeks
  Single limb balance with eyes open and eye closed conditions will be assessed using a Tekscan pressure mat
Change from Baseline Strength | Baseline, 4 weeks
  Ankle and hip strength will be assessed using a handheld dynamometer in N
Change from Baseline Foot and Ankle Ability Measure (FAAM) | Baseline, 4 weeks
  The Foot and Ankle Ability Measure (FAAM) for Activities of Daily Living total score will be assessed. The score will be assessed as a percentage. Scores closer to 100% indicate full ankle function. Lower percentage scores indicate ankle dysfunction.
Change from Baseline Foot and Ankle Ability Measure (FAAM) Sport | Baseline, 4 weeks
  The Foot and Ankle Ability Measure (FAAM) Sport total score will be assessed. The score will be assessed as a percentage. Scores closer to 100% indicate full ankle function. Lower percentage scores indicate ankle dysfunction.
Change from Baseline Identification of Functional Ankle Instability (IdFAI) | Baseline, 4 weeks
  The Identification of Functional Ankle Instability (IdFAI) total score will be assessed. Raw scores will be assessed. Higher scores indicate more ankle dysfunction. Lower scores indicate better ankle function.
Change from Baseline International Physical Activity Questionnaire | Baseline, 4 weeks
  The International Physical Activity Questionnaire total score will be assessed. Higher scores represent increased physical activity.
Change from Baseline Tampa Scale if Kinesiophobia (TSK) | Baseline, 4 weeks
  The Tampa Scale if Kinesiophobia (TSK) total score will be assessed. Lower scores indicate less kinesiophobia. Higher scores indicate higher amount of kinesiophobia.
Change from Baseline Visual Analog Scale (VAS) | Baseline, 4 weeks
  The Visual Analog Scale (VAS) total score will be assessed. The range will be from 0 to 100. Higher score indicates worse ankle pain. Lower score indicates better ankle pain.
The Global Rating of Change (GROC) Score | 4 weeks
  The Global Rating of Change (GROC) score will be assessed at the follow-up visit. A positive and higher score indicates the patient feels better than they did when they began the study. A score of 0 indicates no change from baseline. A negative and lower score indicates the patient feels worse than they did when they began the study.
Change from Baseline Physical Activity | Baseline, 4 weeks
  Fitbit Charge HR monitors will be worn by all participants for 4 weeks. Average daily steps will be analyzed.

CONTACTS AND LOCATIONS:
Overall Officials: Jay N Hertel, PhD, Principal Investigator — University of Virginia
Locations (1):
- University of Virginia, Charlottesville, Virginia, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Waterman BR, Owens BD, Davey S, Zacchilli MA, Belmont PJ Jr. The epidemiology of ankle sprains in the United States. J Bone Joint Surg Am. 2010 Oct 6;92(13):2279-84. doi: 10.2106/JBJS.I.01537. PMID 20926721
- [Background] Delahunt E, Coughlan GF, Caulfield B, Nightingale EJ, Lin CW, Hiller CE. Inclusion criteria when investigating insufficiencies in chronic ankle instability. Med Sci Sports Exerc. 2010 Nov;42(11):2106-21. doi: 10.1249/MSS.0b013e3181de7a8a. PMID 20351590
- [Background] Mok KM, Fong DT, Krosshaug T, Engebretsen L, Hung AS, Yung PS, Chan KM. Kinematics analysis of ankle inversion ligamentous sprain injuries in sports: 2 cases during the 2008 Beijing Olympics. Am J Sports Med. 2011 Jul;39(7):1548-52. doi: 10.1177/0363546511399384. Epub 2011 Apr 1. No abstract available. PMID 21460069
- [Background] Fong DT, Ha SC, Mok KM, Chan CW, Chan KM. Kinematics analysis of ankle inversion ligamentous sprain injuries in sports: five cases from televised tennis competitions. Am J Sports Med. 2012 Nov;40(11):2627-32. doi: 10.1177/0363546512458259. Epub 2012 Sep 11. PMID 22967824
- [Background] Bonnel F, Toullec E, Mabit C, Tourne Y; Sofcot. Chronic ankle instability: biomechanics and pathomechanics of ligaments injury and associated lesions. Orthop Traumatol Surg Res. 2010 Jun;96(4):424-32. doi: 10.1016/j.otsr.2010.04.003. Epub 2010 May 20. PMID 20493797
- [Background] Chinn L, Dicharry J, Hertel J. Ankle kinematics of individuals with chronic ankle instability while walking and jogging on a treadmill in shoes. Phys Ther Sport. 2013 Nov;14(4):232-9. doi: 10.1016/j.ptsp.2012.10.001. Epub 2013 Apr 25. PMID 23623243
- [Background] Doherty C, Bleakley C, Hertel J, Caulfield B, Ryan J, Delahunt E. Recovery From a First-Time Lateral Ankle Sprain and the Predictors of Chronic Ankle Instability: A Prospective Cohort Analysis. Am J Sports Med. 2016 Apr;44(4):995-1003. doi: 10.1177/0363546516628870. Epub 2016 Feb 24. PMID 26912285
- [Background] Donovan L, Hart JM, Saliba SA, Park J, Feger MA, Herb CC, Hertel J. Rehabilitation for Chronic Ankle Instability With or Without Destabilization Devices: A Randomized Controlled Trial. J Athl Train. 2016 Mar;51(3):233-51. doi: 10.4085/1062-6050-51.3.09. Epub 2016 Mar 2. PMID 26934211
- [Background] Donovan L, Hart JM, Saliba S, Park J, Feger MA, Herb CC, Hertel J. Effects of ankle destabilization devices and rehabilitation on gait biomechanics in chronic ankle instability patients: A randomized controlled trial. Phys Ther Sport. 2016 Sep;21:46-56. doi: 10.1016/j.ptsp.2016.02.006. Epub 2016 Feb 27. PMID 27428534
- [Background] Donovan L, Hertel J. A new paradigm for rehabilitation of patients with chronic ankle instability. Phys Sportsmed. 2012 Nov;40(4):41-51. doi: 10.3810/psm.2012.11.1987. PMID 23306414
- [Background] Feger MA, Hertel J. Surface electromyography and plantar pressure changes with novel gait training device in participants with chronic ankle instability. Clin Biomech (Bristol). 2016 Aug;37:117-124. doi: 10.1016/j.clinbiomech.2016.07.002. Epub 2016 Jul 7. PMID 27423026
- [Background] Donovan L, Feger MA, Hart JM, Saliba S, Park J, Hertel J. Effects of an auditory biofeedback device on plantar pressure in patients with chronic ankle instability. Gait Posture. 2016 Feb;44:29-36. doi: 10.1016/j.gaitpost.2015.10.013. Epub 2015 Oct 27. PMID 27004629
- [Background] Koldenhoven RM, Feger MA, Fraser JJ, Saliba S, Hertel J. Surface electromyography and plantar pressure during walking in young adults with chronic ankle instability. Knee Surg Sports Traumatol Arthrosc. 2016 Apr;24(4):1060-70. doi: 10.1007/s00167-016-4015-3. Epub 2016 Feb 8. PMID 26856315
- [Background] Doherty C, Bleakley C, Hertel J, Caulfield B, Ryan J, Delahunt E. Locomotive biomechanics in persons with chronic ankle instability and lateral ankle sprain copers. J Sci Med Sport. 2016 Jul;19(7):524-30. doi: 10.1016/j.jsams.2015.07.010. Epub 2015 Jul 10. PMID 26296816
- [Background] Noehren B, Scholz J, Davis I. The effect of real-time gait retraining on hip kinematics, pain and function in subjects with patellofemoral pain syndrome. Br J Sports Med. 2011 Jul;45(9):691-6. doi: 10.1136/bjsm.2009.069112. Epub 2010 Jun 28. PMID 20584755
- [Background] McKeon PO, Paolini G, Ingersoll CD, Kerrigan DC, Saliba EN, Bennett BC, Hertel J. Effects of balance training on gait parameters in patients with chronic ankle instability: a randomized controlled trial. Clin Rehabil. 2009 Jul;23(7):609-21. doi: 10.1177/0269215509102954. Epub 2009 May 15. PMID 19447844
- [Background] Davis IS, Futrell E. Gait Retraining: Altering the Fingerprint of Gait. Phys Med Rehabil Clin N Am. 2016 Feb;27(1):339-55. doi: 10.1016/j.pmr.2015.09.002. PMID 26616188